CLINICAL TRIAL: NCT05189470
Title: Inforatio Technique to Promote Wound Healing of Diabetic Foot Ulcers: a Parallel-group, Evaluator-blinded, Randomized Clinical Trial
Brief Title: Inforatio Technique to Promote Wound Healing of Diabetic Foot Ulcers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMN-2021-08362; SJ-904 (Other: The Region Zealand Committee on Health Research Ethics); REG-116-2021 (Other: The Region Zealand Research Registry)
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Foot Ulcer; Diabetes; Foot Ulcer; Diabetic Foot; Diabetes Complications; Diabetes Mellitus
Keywords: Diabetic Foot Ulcer; Wound treatment; Inforatio technique
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Healing is assessed on digital ulcer images by assessors that are blinded to treatment allocation. The digital images will be blinded by the primary investigator before delivery to the assessors. Data analysts will also be blinded to treatment allocation. It is not possible to blind participants or the staff that perform wound care and clinical assessment of healing because inforatios are visible in the wound bed after application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): These participants will receive the usual care of the respective outpatient clinics.
  Interventions: Other: Usual care of the respective outpatient clinics
- Intervention group (Experimental): Participants that are randomized to the intervention group will receive both inforatio technique and usual care. Inforatio technique will be applied at baseline, 3, 6, 9 and 12 week- follow-up as long as the ulcers have a diameter of minimum four mms and have not developed infection, necrosis, positive probe-to-bone test, exposure of joint or tendon; or underlying osteomyelitis. In addition, inforatio technique will not be applied on ulcers that are covered by scab if the wound care staff assess that the scab should not be removed from the ulcer.
  Interventions: Procedure: Inforatio technique; Other: Usual care of the respective outpatient clinics

INTERVENTIONS:
Procedure: Inforatio technique — Inforatio technique is a novel minimal invasive procedure where small cuts are made on wound beds with punch biopsy tools near the wound edges but without involving wound edge epithelia. Inforatio technique is applied after the wound has been surgically debrided for slough and devitalized tissue.
  Arms: Intervention group
Other: Usual care of the respective outpatient clinics — Usual care of the DFUs includes local wound care and offloading treatment.

SUMMARY:
This randomized clinical trial will examine the effect of inforatio technique on healing of diabetic foot ulcers (DFUs).

Inforatio technique is a novel procedure developed by the research group. The definition of inforatio technique is application of small cuts in wound beds with punch biopsy tools without involving surrounding epithelia. The aim is to initiate an acute inflammatory response that will promote healing of the ulcers.

DETAILED DESCRIPTION:
BACKGROUND

15-25% of diabetic patients develop chronic foot ulcers - a serious comorbidity that widely affects quality of life and is associated with increased mortality and morbidity. 50-60% of DFUs become infected, and 20% of patients with infected DFUs undergo lower extremity amputation.

Inforatio technique is a novel treatment of DFUs where small cuts are made in wound beds with punch biopsy tools without involving epithelia. The aim is to cause controlled bleeding and initiate an acute inflammatory response that may promote healing.

The research group has conducted a preceding feasibility trial that showed promising results (see study by Moeini et al. in the reference list). Inforatio technique may become a supplemental treatment option for diabetic patients worldwide if it shows a beneficial effect on healing.

TRIAL AIMS

This trial aims to assess whether the proportion of ulcers that heal within 20 weeks is higher when DFUs are treated with inforatio technique in addition to usual wound care compared to treatment with usual wound care alone.

RECRUITMENT

Patients are eligibility-screened and identified by the investigators and wound care staff when patients visit the recruiting wound outpatient clinics.

INCLUSION AND FOLLOW-UP

Eligible patients are included if they give their oral and written consent to participate. The baseline trial visit takes place on the day that patients give their consent to participate.

The trial comprises a 20-week clinical follow-up. Follow-up visits will be at 3, 6, 9, 12, 16 and 20 weeks after baseline (give or take 7 days for midtrial visits and from 20 to 22 weeks after baseline for the last trial visit).

Follow-up end whenever the following appears; 20-week follow-up visit, death, amputation, or the outpatient clinic staff observes healing.

The trial will be stopped if the intervention shows an unintended effect or potential harm.

RANDOMIZATION

Allocation of participants is conducted by block randomization with stratification by center and will be generated with Research Electronic Data Capture (REDCap)©. Block sizes will be randomly alternating between two and four. The allocation will immediately be revealed to the participant and wound care staff. Adequate allocation concealment is ensured by the irreversibility of randomization and the inability to predict the next allocation assignment in RedCap.

STATISTICAL ANALYSIS PLAN

Baseline characteristics will be reported with appropriate descriptive statistics. The analyses of primary and secondary outcomes will be performed on the intention-to-treat population with participants being analyzed as randomized regardless of the treatment received. Supplementary analyses will be performed on the per-protocol population, which excludes participants with one or more serious protocol violations as defined below:

* Participants not receiving their allocated treatment.
* Participants with inadequate adherence, which is defined as the following:

  * Participants that miss more than 3 of the 6 follow-up trial visits.
  * Participants in the intervention group that miss more than 2 of the 4 trial visits where inforatio is applied.

The primary analysis of the trial will be a logistic regression for proportion of healed ulcers with adjustment for center of recruitment.

EQ-5D-5L and Wound-QoL data will be presented descriptively in line with the guidelines for the questionnaires. A multivariate linear regression adjusting for baseline score will be performed for analysis of change in EQ-5D-5L index score and Wound-QoL global score.

Safety outcome will be descriptively reported and analyzed on 'as treated' basis where participants are grouped according to whether they received inforatio technique. Mean time and range from the last inforatio applied to an event is detected will be reported for the intervention group. A statistical comparison between groups will be conducted by chi square test and estimates of relative risk with 95% confidence interval. Inforatio-related adverse events will be descriptively reported.

An interim analyses will be performed after 50 participant has completed follow-up.

Significance is set at p-value <0.05 and p-values are two-tailed. Underlying statistical assumptions for linear and logistic regressions will be assessed graphically.

HANDLING OF MISSING DATA

Data on Wound-QoL global score that is missing due to death during follow-up, will not be considered in the handling of missing data. Otherwise, missing data on primary and secondary outcomes will be handled according to recommendations by Jakobsen et al. (see reference list). If the proportion of missing data on an outcome is <5%, the primary analysis of missing data will be complete-case analyses. If more than 5% data of an outcome is missing, the primary analysis will include missing data imputed by multiple imputation technique and complete case analysis will be performed as a sensitivity analysis. In both cases, a best-worst and worst-best case analysis will be conducted for missing data on healing.

SAMPLE SIZE

A meta analysis by Margolis et al. (see reference list) has reported a healing rate of 30.9% (95% CI 26.6-35.1) in 20 weeks for non-infected DFUs that were treated with standard wound care. A healing rate of 60% in 20 weeks was suggested by the preceding feasibility trial when patients receive inforatio technique in addition to usual wound care.

When the power is 80% and the alpha-level is 5%, a power calculation gives a sample size of 84 for comparison of two proportions when the outcome proportion is 30% for the control group and the aim is to assess whether the outcome improves with 30 percentage points in the intervention group. To allow an attrition of 20%, the aim is to recruit 100 participants for the trial.

ETHICAL CONSIDERATIONS AND RISK ASSESSMENT OF SIDE EFFECTS

Inforatio technique is a minimal invasive procedure. Thus, no adverse events are expected as a result of inforatio technique except from a low risk of pain during application. In the preceding feasibility trial, no intervention-related adverse events were observed and participants did not experience pain during application. Furthermore, inforatio technique showed a promising effect on healing.

The clinical assessment of the wound care staff, patient preference and patient tolerance is taken into consideration before inforatio technique is applied.

If the inforatio technique shows a significant positive effect on healing, it would become of great importance for future patients as a supplemental treatment to standard wound care of DFUs.

COMPETING INTERESTS

The trial investigators declare that they have no competing interests.

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥ 18 years
* Diabetes mellitus
* Non-surgical ulcer located distal to the malleoli
* Wound diameter >4 millimeters
* Patient-reported wound duration ≥ 6 weeks

Only one ulcer will be included from each participant. If a patient has more than one eligible ulcer, the largest ulcer is included. In case of equally sized ulcers, the ulcer with the most recent onset is included.

EXCLUSION CRITERIA

* Dementia or other reasons that cause inability to give informed consent
* Malignant disease
* Current treatment with systemic immunosuppressive drugs.

Exclusion criteria related to the index extremity:

* Diagnosed with or awaiting evaluation of suspected acute phase Charcot arthropathy or osteomyelitis
* Non-palpable pulse in both arteria dorsalis pedis and arteria tibialis posterior accompanied by systolic toe pressure <30 mmHg in the index foot.
* Amputation at midfoot level or proximal to midfoot level
* Revascularization procedure awaits or has been undertaken within the last 8 weeks or the patient awaits a vascular surgeons' decision on revascularization
* Gangrene

Exclusion criteria related to the index ulcer

* Infection of the ulcer defined according to IWGDF/IDSA (International Working Group on the Diabetic Foot/ Infectious Diseases Society of America system) classification as presence of at least 2 of the following; 1) local swelling or induration; 2) erythema >0.5 to ≤2 cm around the ulcer; 3) local tenderness or pain; 4) local warmth; or 5) purulent discharge. Current antibiotic treatment due to infection of the index ulcer will also be considered as an ongoing infection regardless of presence of clinical signs of infection.
* Positive probe-to-bone test
* Exposed joint or tendon
* The soft tissue layer covering bone or joint is evaluated to be too thin to allow for inforatio technique anywhere in the wound bed.
* Interdigital ulcer location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Complete healing | 20 weeks
  Healing is defined as complete epithelialization without any discharge from the site of the index ulcer.
  The primary outcome is the proportion of ulcers in each allocation group where healing is observed based on blinded assessment of digital images from the participants' last trial visit. The assessment of healing on digital images will be performed separately by two blinded assessors. Digital images where disagreement occurs are discussed between the assessors until agreement is reached. Any inconsistencies between the blinded assessment of healing on images and unblinded clinical assessment at trial visits will be reported.
  In case of death and amputation the primary outcome is registered as non-healing.

SECONDARY OUTCOMES:
Change in EQ-5D-5L visual analog scale (EQ VAS) score from baseline to end of follow-up | 20 weeks
  The EQ VAS score is used to assess change in participant-rated health from baseline to end of follow-up.
  Participants fill out the Danish version of the EQ-5D-5L questionnaire at baseline and the last trial visit or after 20 weeks from the day of amputation if participants undergo amputation of their index limb during follow-up. EQ-5D-5L is a general health patient-reported outcome measure that includes a visual analog scale and a descriptive 5-dimension system. Permission to use EQ5-5D-5L (registration ID 39403) has been obtained.
  In case of death, the EQ VAS score will be registered as missing.
Change in Wound-QoL global score from baseline to end of follow-up | 20 weeks
  Wound-QoL global score is used to assess change in disease-specific quality of life from baseline to end of follow-up.
  Participants fill out the Danish version of the Wound-QoL questionnaire at baseline and the last trial visit. The Wound-QoL is a disease-specific patient-reported outcome measure that consists of 17 items, which each has a score from 0 to 4 - 0 indicates no problem and 4 is the highest score for an ulcer-related problem. The global Wound-QoL score is an average of all item scores. In case of death, the Wound-Qol score will be registered as missing. In case of amputation of the index extremity, the Wound-QoL global score is 4, which represents the worst possible outcome for Wound-QoL. The Wound-QoL response is defined as missing if less than 13 of the 17 items have been completed. Permission to the Danish version of the Wound-QoL has been obtained.

OTHER OUTCOMES:
Inforatio related adverse events | 20 weeks
  Inforatio-related adverse events will be descriptively reported. Relatedness to inforatio technique will be qualitatively assessed as definitely related, probably related, probably not, or definitely not related. An event is assessed as probably not related to inforatio technique when the event is most likely to be explained by side effects from other treatments; a natural course of DFUs; or the clinical condition of the participant.
Ulcer-related adverse events | 20 weeks
  Following adverse events related to the index ulcer will be reported:
  * Total wound area increase during follow-up
  * Infection of the ulcer
  * Exposure of bone, tendon or joint in the wound bed
  * Osteomyelitis of underlying bone is diagnosed
  * Surgical wound intervention of the ulcer in an operating theater
  * Hospitalization related to the ulcer
  * Minor amputation of the index extremity (below ankle)
  * Major amputation of the index extremity (above ankle)
  * Mortality related to the ulcer
  The events will be descriptively reported and analyzed on 'as treated' basis where participants are grouped according to whether they received inforatio technique. Mean time and range from the last inforatio applied to an event is detected will be reported for the intervention group. A statistical comparison between groups will be conducted for proportion of participants experiencing one or more adverse events related to the index ulcer.
Patient-reported adverse events | 20 weeks
  * Patient-reported adverse events related to index ulcers: Participants are asked at each follow-up visit whether they have experienced onset of an ulcer-related adverse events since their last trial visit.
  * Adverse events related to inforatio technique application: Participants from the intervention group are asked after each inforatio technique application whether they experience any adverse events during or immediately after application.
Serious adverse events | 20 weeks
  Serious adverse events are defined according to FDA (U.S. Food and Drug Administration) as death, life-threatening events, hospitalization, disability or permanent damage. The outcome will be descriptively reported and analyzed on 'as treated' basis where participants are grouped according to whether they received inforatio technique. A statistical comparison between groups will be conducted for proportion of serious adverse events.
One-year mortality | 1 year
  Events of death during the first year from baseline.
One-year amputation rate | 1 year
  Events of amputation in index extremities during the first year from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Moeini, MD, Principal Investigator — Zealand University Hospital; Hans Gottlieb, MD PhD, Study Chair — University of Copenhagen; Tue S Jørgensen, MD PhD, Study Chair — Zealand University Hospital; Thomas V Aagaard, PT MsC, Study Chair — Holbaek Hospital; Maj R Kornø, MD, Study Chair — Nykoebing Falster Hospital; Malene RB Larsen, MD, Study Chair — Zealand University Hospital; Stig Brorson, MD PhD DMsc, Principal Investigator — Zealand University Hospital
Locations (4):
- Denmark (4):
  - Herlev University Hospital, Department of Orthopaedic Surgery, Herlev
  - Zealand University Hospital, Department of Orthopaedic Surgery, Køge
  - Nykoebing Falster Hospital, Nykøbing Falster
  - Slagelse Hospital, Department of Orthopaedic Surgery, Slagelse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews KL, Houdek MT, Kiemele LJ. Wound management of chronic diabetic foot ulcers: from the basics to regenerative medicine. Prosthet Orthot Int. 2015 Feb;39(1):29-39. doi: 10.1177/0309364614534296. PMID 25614499
- [Background] Karri VV, Kuppusamy G, Talluri SV, Yamjala K, Mannemala SS, Malayandi R. Current and emerging therapies in the management of diabetic foot ulcers. Curr Med Res Opin. 2016;32(3):519-42. doi: 10.1185/03007995.2015.1128888. Epub 2016 Jan 12. PMID 26643047
- [Background] Zimny S, Pfohl M. Healing times and prediction of wound healing in neuropathic diabetic foot ulcers: a prospective study. Exp Clin Endocrinol Diabetes. 2005 Feb;113(2):90-3. doi: 10.1055/s-2004-830537. PMID 15772900
- [Background] Greer N, Foman NA, MacDonald R, Dorrian J, Fitzgerald P, Rutks I, Wilt TJ. Advanced wound care therapies for nonhealing diabetic, venous, and arterial ulcers: a systematic review. Ann Intern Med. 2013 Oct 15;159(8):532-42. doi: 10.7326/0003-4819-159-8-201310150-00006. PMID 24126647
- [Background] Devlin N, Parkin D, Janssen B. Methods for Analysing and Reporting EQ-5D Data [Internet]. Cham (CH): Springer; 2020. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK565678/ PMID 33347096
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Margolis DJ, Kantor J, Berlin JA. Healing of diabetic neuropathic foot ulcers receiving standard treatment. A meta-analysis. Diabetes Care. 1999 May;22(5):692-5. doi: 10.2337/diacare.22.5.692. PMID 10332667
- [Background] Moeini S, Gottlieb H, Jorgensen TS, Larsen MRB, Brorson S. Treatment of Diabetic Foot Ulcers With Inforatio Technique to Promote Wound Healing: A Feasibility Trial. Int J Low Extrem Wounds. 2023 Jun;22(2):241-250. doi: 10.1177/15347346211002364. Epub 2021 Apr 28. PMID 33909504
- [Background] Monteiro-Soares M, Russell D, Boyko EJ, Jeffcoate W, Mills JL, Morbach S, Game F; International Working Group on the Diabetic Foot (IWGDF). Guidelines on the classification of diabetic foot ulcers (IWGDF 2019). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3273. doi: 10.1002/dmrr.3273. PMID 32176445
- [Derived] Moeini S, Gottlieb H, Jorgensen TS, Aagaard TV, Korno MR, Larsen MRB, Brorson S. Inforatio technique to promote wound healing of diabetic foot ulcers: study protocol for a parallel-group, evaluator-blinded, randomised clinical trial. BMJ Open. 2022 Sep 19;12(9):e062344. doi: 10.1136/bmjopen-2022-062344. PMID 36123051
- See also: Chadwick P, Edmonds M, Mccardle J, Armstrong D. International Best Practice Guidelines: Wound management in diabetic foot ulcers. Wounds International. Published 2013. Accessed November 26, 2020. — http://www.woundsinternational.com/resources/details/best-practice-guidelines-wound-management-diabetic-foot-ulcers
- See also: EuroQol Research Foundation. EQ-5D-5L User Guide. Published 2019. Accessed December 16, 2020. — http://euroqol.org/publications/user-guides/
- See also: Wound-QoL. Wound-QoL User Manual. User Manual for the questionnaire on quality of life with chronic wounds. Published 2020. Accessed January 20, 2021. — http://www.wound-qol.com/download/
- See also: FDA. What is a Serious Adverse Event? Published 2016. Accessed December 16, 2020. — http://www.fda.gov/safety/reporting-serious-problems-fda/what-serious-adverse-event